CLINICAL TRIAL: NCT01885520
Title: A Randomized,Open-label, Single-dose, Crossover Clinical Trial to Evaluate the Food Effect on the Pharmacokinetics of Eperisone HCl SR Tablet 75mg After Oral Administration in Healthy Adult Male Subjects.
Brief Title: Clinical Trial to Evaluate the Food Effect on the Pharmacokinetics of Eperisone HCl SR Tablet 75mg
Acronym: eperisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NVP-EPT-PK-02
Record Dates: First submitted 2013-06-15; First posted 2013-06-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Low Back Pain
Keywords: low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fasting condition (Experimental): eperisone SR administrated under fasting condition
  Interventions: Dietary Supplement: fasting condition
- Fed condition (Active Comparator): eperisone SR administrated under fed condition
  Interventions: Dietary Supplement: fed condition

INTERVENTIONS:
Dietary Supplement: fasting condition — eperisone SR tablet 75mg administrated under fasting
  Arms: fasting condition
Dietary Supplement: fed condition — eperisone SR tablet 75mg administrated fed condition
  Arms: Fed condition

SUMMARY:
The purpose of this study is to evaluate the food effect on the pharmacokinetics of eperisone HCl SR tablet

DETAILED DESCRIPTION:
eperisone hydrochloride(muscle relaxant)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age between 20 and 55 signed informed consent

Exclusion Criteria:

* Hypotension or hypertension has a history of allergy reaction of this drug or other drugs

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
AUC | 0-24h
Cmax | 0-24h

SECONDARY OUTCOMES:
T1/2 | 0-24h
Tmax | 0-24h

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Yo Ran, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Jung-gu, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No